CLINICAL TRIAL: NCT06248619
Title: A Phase 3, Randomized, Double-masked, Placebo-controlled, Parallel-group, Multicenter Trial to Evaluate the Efficacy, Safety and Tolerability of Subcutaneous Teprotumumab in Participants With Moderate-to-Severe Active Thyroid Eye Disease
Brief Title: A Trial to Investigate Teprotumumab Subcutaneous Administration Compared With Placebo in Male and Female Adult Participants With Moderate-to-severe Active Thyroid Eye Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZNP-TEP-305
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
Keywords: Teprotumumab; Active Thyroid Eye Disease; Tepezza; Teprotumumab-trbw
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teprotumumab (Experimental): Teprotumumab administered SC
  Interventions: Biological: Teprotumumab
- Placebo (Placebo Comparator): Placebo for teprotumumab administered SC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Teprotumumab — SC injection
  Arms: Teprotumumab
Other: Placebo — SC injection
  Arms: Placebo

SUMMARY:
The study consists of a randomized double-masked, placebo-controlled, parallel-group, multicenter trial with an optional open-label treatment period for proptosis non-responders who complete the Double-masked Treatment Period.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effect of teprotumumab subcutaneous administration versus placebo on the proptosis responder rate (ie, the percentage of participants with a ≥ 2-mm reduction from Baseline in the study eye without deterioration [≥ 2-mm increase] of proptosis in the fellow eye) at Week 24.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide written informed consent.
2. Participant can be male or female and must be between the ages of 18 and 80 years, inclusive, at Screening.
3. Participant must have a clinical diagnosis of Graves' disease associated with active TED with a CAS ≥ 3 (on the 7-item scale) for the most severely affected eye at Screening and Baseline.
4. Participant must have moderate-to-severe active TED (not sight-threatening but has an appreciable impact on daily life), usually associated with 1 or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement and/or inconstant or constant diplopia. (Note: Participants with no diplopia at Baseline will be limited to approximately 25% of the total number enrolled.)
5. Participant has proptosis ≥ 3 mm from Baseline (prior to diagnosis of TED), as estimated by treating physician, and/or proptosis ≥ 3 mm above normal for race and gender.
6. Participant had onset of active TED symptoms (as determined by participant records) within 15 months prior to Baseline.
7. Participants must be euthyroid with the baseline disease under control or have mild hypoor hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine [FT3] levels < 50% above or below the normal limits) at Screening. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of the trial.
8. Participant does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the trial.
9. Women of childbearing potential must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified time points (ie, prior to each dose and throughout participation in the trial).
10. Participant is willing and able to comply with the protocol requirements for the duration of the trial.

Exclusion Criteria:

1. Participant has decreased best-corrected visual acuity due to optic neuropathy, defined by a decrease in vision of 2 lines on the Snellen chart (or equivalent), new visual field defect or color defect secondary to optic nerve involvement within the last 6 months.
2. Participant has corneal decompensation unresponsive to medical management.
3. Participant has a decrease in CAS of ≥ 2 points between Screening and Baseline.
4. Participant has a decrease in proptosis of ≥ 2 mm between Screening and Baseline.
5. Participant had prior orbital irradiation, orbital decompression or strabismus surgery (excluding childhood strabismus surgeries unrelated to TED/Graves' disease).
6. Participant is planning to have eyelid surgery during the trial.
7. Participant received periocular botulinum toxin injection within 12 months prior to Screening.
8. Participant has any systemic use of a steroid (IV or oral) or steroid eye drops for the treatment of TED or other conditions within 3 weeks prior to Screening. Exceptions include local administration (excluding periocular), eg, topical, intra-articular, and inhaled steroids, as well as steroids used to treat infusion reactions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Proptosis responder rate (percentage of participants with a ≥ 2-mm reduction from baseline in proptosis in the study eye without deterioration [≥ 2-mm increase] of proptosis in the fellow eye). | Week 24

SECONDARY OUTCOMES:
Mean change from Baseline in proptosis measurement in the study eye | Week 24
Overall responder rate (percentage of participants with ≥ 2-point reduction in CAS AND ≥ 2-mm reduction in proptosis from Baseline, provided there is no corresponding deterioration [≥ 2-point/mm increase] in CAS or proptosis in the fellow eye) | Week 24
Percentage of participants with a CAS value of 0 or 1 | Week 24
Change from Baseline in diplopia as ordinal response categories | Week 24
Diplopia responder rate, defined as the percentage of participants with Baseline binocular diplopia > 0 who have a reduction of ≥ 1 grade | Week 24
Complete diplopia responder rate, defined as the percentage of participants with a Baseline binocular diplopia score > 0 and a score of 0 | Week 24
Mean change from Baseline in the GO-QoL questionnaire overall score | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- United States (11):
  - Catalina Eye Care - NVISION - PPDS, Tucson, Arizona
  - Advanced Quality Medical Research, Orland Park, Illinois
  - W Kellogg Eye Center, Ann Arbor, Michigan
  - Las Vegas Endocrinology, Henderson, Nevada
  - The Center for Eye and Facial Plastic Surgery, Somerset, New Jersey
  - Casey Eye Institute -515 SW Campus Dr, Portland, Oregon
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center - 848 Adams Ave, Memphis, Tennessee
  - Baylor College of Medicine-1977 Butler Blvd, Houston, Texas
  - University of Washington Eye Institute, Seattle, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Argentina (3):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Organización Médica de Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Medico Grupo Laser Vision, Rosario, Santa Fe Province
- Australia (4):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Queensland Eye Institute, Wooloongabba, Queensland
  - Royal Adelaide Hospital, Adelaie, South Australia
  - Centre For Eye Research Australia Ltd, East Melbourne, Victoria
- Canada (3):
  - Vancouver Coastal Health Research Institute (VCHRI) - 2550 Willow St, Vancouver, British Columbia
  - McGill University Health Centre Research Institute, Montreal, Quebec
  - CHU de Quebec-Universite Laval CUO Recherche Clinique Hopital du St-Sacrement, Québec
- AP-HM-Hôpital de La Conception, Marseille, Bouches-du-Rhône, France
- Universitätsklinikum Essen, Essen, North Rhine-Westphalia, Germany
- Italy (3):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa
- Japan (5):
  - Hayashi Eye Hospital, Fukuoka, Hukuoka
  - Kozawa Eye hospital and Diabetes Center, Mito, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Gokeikai Osaka Kaisei Hospital, Osaka-Shi Yodogawa-Ku, Ôsaka
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia-Avda de Fernando Abril Martorell 106, Valencia
- Taiwan (3):
  - Changhua Christian Hospital, Changhua County
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Moorfields Eye Hospital - PPDS, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com